CLINICAL TRIAL: NCT02277327
Title: Randomized Controlled Trial to Decrease Admission Rates in Medically Complex Children in a Medical Home Program
Brief Title: Trial to Reduce Hospitalizations in Children With Medical Complexity
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Thomas Klitzner, MD, PhD, Executive Directior, Pediatric Medical Home Program at UCLA, University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: UCLAMedHomeRCT
Record Dates: First submitted 2014-10-24; First posted 2014-10-29 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Chronic Illness
Keywords: Hospitalization; Readmissions; Medical complexity
MeSH Terms: conditions — Chronic Disease | interventions — Patient Transfer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Subjects randomized to the "intervention group" will participate in a bundled intervention that includes action planning and care transitions (for those hospitalized during the study period)
  Interventions: Behavioral: Plans of Action and Care Transitions
- Routine Care (Placebo Comparator): Subjects randomized to the "routine care" group will continue to receive their usual care from the Pediatric Medical Home Program at UCLA
  Interventions: Behavioral: Routine Care

INTERVENTIONS:
Behavioral: Plans of Action and Care Transitions — Subjects randomized to the "intervention" will participate in action planning and care transitions (if hospitalized during the study period)
  Arms: Intervention
Behavioral: Routine Care — Subjects randomized to the "control" group will continue to receive routine care within the medical home program
  Arms: Routine Care

SUMMARY:
The investigators hypothesize that an intervention, within an established patient-centered medical home, aimed at reducing modifiable risks for hospitalization, can decrease hospital utilization among medically complex children.

DETAILED DESCRIPTION:
The investigators will pilot test an intervention that includes contingency planning and care transitions within an established medical home program caring for children with medical complexity. Children with medical complexity receiving care within the UCLA Medical Home Program will be randomized to the pilot intervention or usual medical home care. The primary goal will be to reduce admissions and readmissions in the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 0 to 17 years old who are enrolled in the Pediatric Medical Home Program at UCLA
* English and Spanish-speaking only

Exclusion Criteria:

* Children older than 17 years old who are enrolled in the Pediatric Medical Home Program
* Non-English and Non-Spanish speakers

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
(1) number of all-cause admissions, defined as any admission occurring during the study period | 18 to 24 months
(2) preventable admissions, defined by 2 independent physicians blinded to study assignment as an admission due primarily to one of the preventable factors identified from Phase 1 of the study | 18 to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Klitzner, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States